CLINICAL TRIAL: NCT06699368
Title: Clinical Study on the Risk of Left Atrial POP Ablation and Esophageal Injury Under Ultra-High Power and Related Influencing Parameters
Acronym: UHP-POP-ESO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hanxiong Liu, Principal Investigator, The Third People's Hospital of Chengdu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDSY-UHP-POP-ESO
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ultra-High Power Ablation,Safety of Atrial Fibrillation Ablation
Keywords: Ultra-High Power Ablation,Safety of Atrial Fibrillation Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ultra-High-Power Ablation Group (Experimental): The ultra-high-power ablation group will use the QDOT ablation catheter with a power of 90W, ablation points at site 3, inter-point distance maintained at 4-5mm, pressure maintained at 5-30g. The cold saline flow rate during ablation is 8ml/min, and the ablation device will adjust power and saline flow rate based on the electrode temperature at the tip of the QDOT ablation catheter. The target temperature is 60°C, and the cut-off temperature is 65°C, with an ablation endpoint of 4 seconds.
  Interventions: Procedure: The ultra-high-power ablation group
- High-Power Ablation Group (Active Comparator): The high-power ablation group will use the STSF ablation catheter with a power of 50W, ablation points at site 3, inter-point distance maintained at 4-5mm, pressure maintained at 5-30g, and a cold saline flow rate of 15ml/min during ablation. The ablation endpoint for the posterior wall of the left atrium is an Ablation Index (AI) value of 360-410, for the anterior wall 450-480, and for the bottom and top of the left atrium 420-450.
  Interventions: Procedure: The high-power ablation group

INTERVENTIONS:
Procedure: The ultra-high-power ablation group — The ultra-high-power ablation group will use the QDOT ablation catheter with a power of 90W, ablation points at site 3, inter-point distance maintained at 4-5mm, pressure maintained at 5-30g. The cold saline flow rate during ablation is 8ml/min, and the ablation device will adjust power and saline flow rate based on the electrode temperature at the tip of the QDOT ablation catheter. The target temperature is 60°C, and the cut-off temperature is 65°C, with an ablation endpoint of 4 seconds.
  Arms: Ultra-High-Power Ablation Group
Procedure: The high-power ablation group — The high-power ablation group will use the STSF ablation catheter with a power of 50W, ablation points at site 3, inter-point distance maintained at 4-5mm, pressure maintained at 5-30g, and a cold saline flow rate of 15ml/min during ablation. The ablation endpoint for the posterior wall of the left atrium is an Ablation Index (AI) value of 360-410, for the anterior wall 450-480, and for the bottom and top of the left atrium 420-450.
  Arms: High-Power Ablation Group

SUMMARY:
This study aims to evaluate the risks of steam pop (POP) and esophageal injury, as well as related influencing parameters, under ultra-high power ablation technology. In the treatment of arrhythmias such as atrial fibrillation, cardiac ablation surgery is a common method. The use of ultra-high power ablation technology can shorten the operation time and improve effectiveness, but it may also increase the risk of damage to surrounding structures such as the esophagus. We will recruit a certain number of patients who are scheduled to undergo ultra-high power ablation surgery. We will record various parameters during the surgery, such as energy, time, and contact force, and monitor patients for signs of esophageal injury after the surgery. We expect that through this study, we can better understand the potential risks of ultra-high power ablation to the esophagus and identify the key parameters affecting these risks. This will help to improve surgical techniques, reduce complications, and enhance patient safety and surgical outcomes.

DETAILED DESCRIPTION:
This study aims to evaluate the risks of steam pop (POP) and esophageal injury, as well as related influencing parameters, under ultra-high power ablation technology. In the treatment of arrhythmias such as atrial fibrillation, cardiac ablation surgery is a common method. The use of ultra-high power ablation technology can shorten the operation time and improve effectiveness, but it may also increase the risk of damage to surrounding structures such as the esophagus. We will recruit a certain number of patients who are scheduled to undergo ultra-high power ablation surgery. We will record various parameters during the surgery, such as energy, time, and contact force, and monitor patients for signs of esophageal injury after the surgery. We expect that through this study, we can better understand the potential risks of ultra-high power ablation to the esophagus and identify the key parameters affecting these risks. This will help to improve surgical techniques, reduce complications, and enhance patient safety and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 80 years old.
2. Diagnosed with drug-refractory, symptomatic, paroxysmal atrial fibrillation.
3. Non-valvular atrial fibrillation.
4. Able to understand the purpose of the study, voluntarily participate in this research, and the patient or their legal representative signs the informed consent form, willing to complete follow-ups as required by the protocol.

Exclusion Criteria:

1. Atrial fibrillation secondary to thyroid disease or other reversible factors;
2. Imaging studies indicating intracardiac thrombus;
3. Moderate to severe mitral stenosis or regurgitation;
4. Left ventricular ejection fraction <40%, or New York Heart Association (NYHA) functional class III or IV;
5. Unstable angina;
6. Myocardial infarction (MI) or coronary artery bypass grafting (CABG) within 3 months prior to enrollment;
7. Presence of mural thrombus, space-occupying disease, or other abnormalities that hinder vascular puncture or catheter manipulation;
8. Contraindications to anticoagulation and a history of blood coagulation or bleeding abnormalities;
9. Patients with active systemic infections; Patients who have had an atrial septal closure device implanted within the last 6 weeks;
10. Female patients who are pregnant, breastfeeding, or unable to use contraception during the study period;
11. Patients with a life expectancy of less than 12 months (e.g., advanced malignant tumors); patients who have had an atrial septal closure device implanted within the last 6 weeks;
12. Conditions affecting vascular access;
13. Patients who are concurrently participating in other drug or device clinical trials;
14. Any other abnormalities or diseases that the investigator deems should exclude the patient from the study enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-28 (Estimated); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
The number of times the esophageal temperature monitoring electrode shows a temperature exceeding 38.5°C | Intraoperative Immediate
  The number of times the esophageal temperature monitoring electrode shows a temperature exceeding 38.5°C

SECONDARY OUTCOMES:
The number of times Intraoperative steam POP occurrence | Intraoperative Immediate
  The number of times Intraoperative steam POP occurrence

OTHER OUTCOMES:
Whether esophageal injury and related complications such as esophageal fistula occur within one month postoperatively | 1 Months Post-Operation
Occurrence of chronic pericardial and POP-related complications within 7 days postoperatively | 7 days Post-Operation.
  Occurrence of chronic pericardial and POP-related complications within 7 days postoperatively

IPD SHARING:
Plan to Share IPD: Undecided